CLINICAL TRIAL: NCT06941948
Title: Prospective Clinical Study Design: the Association of Sleep Disorders With Tumor Immune Microenvironment and Prognosis of Lung Cancer
Brief Title: Sleep Disorders and Tumor Immune Microenvironment
Status: Recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-4-17-SD-lung-prospect
Record Dates: First submitted 2025-04-16; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Impact of Sleep Disorders on Tumor Immune Microenvironment and Clinical Outcomes in Lung Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lung cancer-no SD
  Interventions: Other: PSQI
- Lung cancer-SD
  Interventions: Other: PSQI

INTERVENTIONS:
Other: PSQI — PSQI

SUMMARY:
Title: Impact of Sleep Disorders on Tumor Immune Microenvironment and Clinical Outcomes in Lung Cancer: A Prospective Cohort Study

Objective:

This prospective study aims to investigate the causal relationship between sleep disorders (e.g., insomnia, obstructive sleep apnea [OSA]) and alterations in the tumor immune microenvironment (TIME) in lung cancer patients, and to evaluate their joint effects on immunotherapy response and long-term prognosis.

Study Design:

Prospective observational cohort study with 3-year follow-up. Participants: Newly diagnosed primary lung cancer patients (NSCLC/SCLC) prior to treatment initiation (n = 400, target sample size*).

Exposure Groups: Stratified by sleep disorder status (confirmed via polysomnography [OSA] and validated questionnaires [e.g., PSQI ≥7 for insomnia]).

DETAILED DESCRIPTION:
1. Background support Sleep disorders are common in patients with lung cancer, and the incidence is as high as 52.6%-70%, which is related to tumor progression and immunosuppression. Animal experiments have shown that circadian rhythm disruption can reshape the tumor microenvironment, suppress immune responses (such as macrophage dysfunction), and lead to accelerated tumor growth.

   o Clinical data show that the immune status of lung cancer patients, such as PD-L1 expression, T cell infiltration level, is closely related to treatment response and survival rate. However, there is still a lack of prospective research evidence on how sleep disorders affect the progression of lung cancer by regulating the immune microenvironment.
2. Scientific hypothesis

It is hypothesized that sleep disorders (e.g., insomnia, circadian rhythm disruption) affect the tumor immune microenvironment of lung cancer patients through the following mechanisms:

* inhibits the activity of anti-tumor immune cells, such as CD8+ T cells and NK cells;
* promotes the infiltration of immunosuppressive cells (e.g., regulatory T cells, M2 macrophages);
* up-regulates the expression of proinflammatory factors (e.g., IL-6, TNF-α) and inhibits immune checkpoints (e.g., PD-L1), thereby accelerating tumor progression and reducing treatment efficacy.

  2. Study design and methods
  1. Study type Prospective cohort study, stratified analysis of sleep disorder group and non-sleep disorder group, followed up for 1-3 years.
  2. Study subjects
* Inclusion criteria: patients with newly diagnosed stage Ⅲ-Ⅳ non-small cell lung cancer (NSCLC) who had not received systemic therapy (chemotherapy, immunotherapy or radiotherapy);
* Exclusion criteria: patients with serious mental illness, other malignant tumors or receiving sleep medication;
* According to the Pittsburgh Sleep Quality Index (PSQI) score, PSQI≥7 were divided into sleep disorder group, PSQI<7 were divided into control group.

  3. Core indicators Indicator categories Specific indicators Sleep assessment PSQI score, polysomnography (total sleep time, sleep efficiency, and number of awakenings) 10 Immunological indicators of peripheral blood: CD4+/CD8+ T cell ratio, NK cell activity, IL-6, TNF-α levels; Tumor tissue: PD-L1 expression, tumor infiltrating lymphocytes (TILs) density, macrophage polarization (M1/M2) Clinical outcomes Time to progression (TTP), overall survival (OS), response rate (ORR) Auxiliary indicators: Anxiety and Depression Scale (HADS), quality of life score (EORTC QLQ-C30) 4. Data collection and follow-up
* Baseline data: demographic characteristics, tumor stage, molecular subtype (e.g., KRAS mutation status).6
* Dynamic monitoring: sleep quality, immune indicators and tumor burden (imaging) were evaluated every 3 months;
* Interventions: Non-pharmacological interventions (e.g., cognitive behavioral therapy, light therapy) 2 were implemented in the sleep-disordered group, and changes in immune indicators were observed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed stage III-IV non-small-cell lung cancer (NSCLC) not receiving systemic therapy (chemotherapy, immunotherapy, or radiotherapy)

Exclusion Criteria:

* Patients with severe mental illness, other malignant tumors, or receiving sleep medication

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study type: Prospective cohort study (single center).
  Data sources:
  Recruitment Organization: Patients with newly diagnosed primary lung cancer (confirmed histopathologically or cytologically) were enrolled at [Zhong shan hospital].
  Time frame: January 2024 to December 2026 (recruitment period).
  Data collection:
  Clinical data: electronic medical record system (EMR), imaging reports, laboratory databases.
  Biological samples: baseline tumor tissue (biopsy/surgical specimens), serial serum/plasma samples (baseline and treatment follow-up time points).
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
TTP | Baseline: Immune indicators assessed at initial diagnosis (pre-treatment)

CONTACTS AND LOCATIONS:
Locations (1):
- Zhong Shan hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No